CLINICAL TRIAL: NCT01491295
Title: Randomized Trial of Switch to Tenofovir Versus Continue Lamivudine/Adefovir Treatment in Lamivudine-resistance Chronic Hepatitis B Patients Who Have Undergone Lamivudine/Adefovir Add-on Treatment
Brief Title: Switch to Tenofovir Versus Continue Lamivudine/Adefovir Treatment in Lamivudine-resistance Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); China Medical University Hospital (Other); Chi Mei Medical Hospital (Other); Chiayi Christian Hospital (Other)
Responsible Party: Principal Investigator, vghtpe user, Professor: Yi-Hsiang Huang, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-174-0194
Record Dates: First submitted 2011-10-27; First posted 2011-12-13 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Hepatitis B
Keywords: Lamivudine; adefovir add on treatment; tenofovir; chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; Lamivudine; adefovir; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamivudine plus adefovir (Active Comparator): Continue lamivudine/adefovir add on treatment (standard treatment)
  Interventions: Drug: Lamivudine plus adefovir
- Tenofovir (Experimental): Switch from lamivudine/adefovir add on threatment to tenofovir monotherapy
  Interventions: Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — Tenofovir disoproxil fumarate 300mg QD for 36 months (adjust dosage according to renal function)
  Other Names: Viread
  Arms: Tenofovir
Drug: Lamivudine plus adefovir — Lamivudine 100mg QD for 36 months (adjust dosage according to renal function) Adefovir 10mg QD for 36 months (adjust dosage according to renal function)
  Other Names: Zeffix; Hepsera
  Arms: Lamivudine plus adefovir

SUMMARY:
1. Adefovir add-on therapy is superior to switching to adefovir monotherapy or entecavir 1mg monotherapy for chronic hepatitis B (CHB) patients with lamivudine resistance (LAM-R)
2. Long-term adefovir add-on therapy was effective for viral suppression. However, the economic burden for such dual antiviral therapy is heavy because of infinite treatment.
3. Tenofovir disoproxil fumarate (TDF) is a potent antiviral agent. TDF demonstrated potent antiviral efficacy in a subset of lamivudine experienced HBeAg-positive patients. TDF is also superior to ADV in HBeAg-negative and HBeAg-positive treatment-naive patients.
4. Theoretically, TDF can replace LAM/ADV when viral suppression has been achieved by LAM/ADV combination treatment in LAM-R CHB patients.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) is a partially double-stranded DNA virus. HBV infection can induce a spectrum of disease ranging from asymptomatic infection to severe chronic liver diseases, including cirrhosis and hepatocellular carcinoma (HCC). Chronic HBV infection is also a major cause of HCC in Taiwan. Over 350 millions people worldwide are chronically infected with HBV. Lamivudine was the first marketing and is the first-line oral anti-viral agent for the therapy of chronic hepatitis B. Infinite nucleoside analogue therapy may be needed for long-term viral suppression especially in patients with HBeAg-negative chronic hepatitis B. The initial randomized studies demonstrated the clinical benefit and safety of lamivudine in both hepatitis B e antigen (HBeAg)-positive and -negative chronic hepatitis B patients. But as high as 20% of the cases under 1-year lamivudine treatment developed genotypic resistance, which defined as the presence of YMDD mutation on the HBV polymerase region. Genotypic resistance is almost always associated with virological breakthrough and exacerbation of liver function. Long-term lamivudine therapy was reported increase HBeAg seroconversion and provided clinical improvement in ALT levels. However, in a four-year follow-up study, YMDD-variant HBV was detected in as high as 67% of patients under lamivudine treatment. Several clinical studies have proven that adefovir add-on therapy is superior to switching to adefovir monotherapy or entecavir 1mg monotherapy for chronic hepatitis B (CHB) patients with lamivudine resistance (LAM-R). Currently, AASLD and EASL guidelines recommend adefovir add-on therapy as a standard treatment for LAM-R CHB patients. Long-term adefovir add-on therapy was effective for viral suppression (8). However, the economic burden for such dual antiviral therapy is heavy because of infinite treatment.

Tenofovir disoproxil fumarate (TDF) is a potent antiviral agent. TDF and ETV are recommended oral first-line therapies for CHB. TDF demonstrated potent antiviral efficacy in a subset of lamivudine experienced HBeAg-positive patients. TDF is also superior to ADV in HBeAg-negative and HBeAg-positive treatment-naive patients. Theoretically, TDF can replace LAM/ADV when viral suppression has been achieved by LAM/ADV combination treatment in LAM-R CHB patients. This clinical trial is a proof of concept study to evaluate the efficacy of switching to TDF monotherapy in such patients.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg-positive for more than 6 months (HBeAg-positive or HBeAg-negative).
* Age > 20 y/o.
* Under lamivudine/adefovir treatment for more than 1 year due to previous lamivudine resistance (LAM-R), current HBV DNA is undetectable (< 20 IU/ml) during enrollment.

Exclusion Criteria:

* HCV, HIV, HDV coinfection.
* Uncontrolled HCC, malignancy or decompensated liver cirrhosis (CTP score ≥ 7).
* Uremia patients or Creatinine ≥ 2 mg/dl.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-09; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of virological breakthrough (defined as HBV DNA > 100 IU/ml) | Sustained viral suppression after switching to TDF for 36 months

SECONDARY OUTCOMES:
HBeAg seroconversion (for HBeAg-positive patients) | HBeAg seroconversion rate at 1, 2 and 3 years
Incidence of HBsAg loss | Incidence of HBsAg loss at 1-, 2-, and 3 -years

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsiang Huang, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital-Division of Gastroenterology, Taipei, Taiwan